CLINICAL TRIAL: NCT02475252
Title: Prospective Case-control Study to Assess the Construct Validity of a Diagnostic Hysteroscopy in a Pelvic Training Model Using an Objective Structured Assessment of Technical Skills (OSATS) Assessment
Brief Title: Construct Validity of a Diagnostic Hysteroscopy Training Model
Acronym: HSK-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment too slow; study completion not possible within frame
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Prof. Clemens Tempfer, MD, Ruhr University of Bochum
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK-2
Record Dates: First submitted 2015-05-03; First posted 2015-06-18 (Estimated); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experts (Active Comparator): Surgically experienced gynecologists with a personal history of at least 50 hysteroscopy procedures will perform a hysteroscopy on a training model.
  Interventions: Procedure: hysteroscopy on a training model
- Novices (Experimental): Medical students will perform a hysteroscopy on a training model.
  Interventions: Procedure: hysteroscopy on a training model

INTERVENTIONS:
Procedure: hysteroscopy on a training model — Diagnostic hysteroscopy on a diagnostic hysteroscopy training model using a pelvic dummy and all surgical instruments also used in the original procedure. The performance of all participants will be scored using an OSATS scoring sheet developed for assessing surgical proficiency.

SUMMARY:
In a prospective case-control study, the investigators compare the Objective Structured Assessment of Technical Skills (OSATS) scores in medical students and gynecologic experts performing a hysteroscopy on a training model for diagnostic hysteroscopy. The investigators hypothesize that OSATS on a hysteroscopy training model has construct validity to discriminate between experts and novices.

DETAILED DESCRIPTION:
In a prospective case-control study, 140 medical students (,novices') and 10 senior gynecologists (,experts') will watch a demonstration detailing how to perform a hysteroscopy on a training model. All probands will perform a hysteroscopy themselves within 1 hour after the demonstration. Their performance will be judged using an Objective Structured Assessment of Technical Skills (OSATS) assessment. Using metrical and non-metrical measurements, construct validity of the hysteroscopy training model to distinguish between experts and novices will be assessed. Secondary endpoints are differences in OSATS scores within the group of novices based on gender and handyness, as well as satisfaction of the novices with the learning experience.

ELIGIBILITY:
Inclusion Criteria:

* medical Student
* no previous experience in gynecologic surgery
* no previous gynecologic surgery Training
* gynecologist with a personal history of at least 50 hysteroscopies)

Exclusion Criteria:

* language barrier
* unwillingness to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Construct validity | within 1 hour after demonstration
  Predefined OSATS scores (metrical and non-metrical items) will be compared between experts and novices

SECONDARY OUTCOMES:
OSATS scores according to gender | within 1 hour after demonstration
  OSATS scores will be compared depending on gender
OSATS scores according to handyness | within 1 hour after demonstration
  OSATS scores will be compared depending on handyness (right- versus left-handed)

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Dept. OBGYN Ruhr University Bochum, Herne, Germany